CLINICAL TRIAL: NCT00854789
Title: Phase Ib Trial of HER2/Neu Peptide (E75) Vaccine in Node Negative Breast Cancer Patients
Brief Title: Safety and Efficacy Study of HER2/Neu (E75) Vaccine in Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: COL George Peoples, MD, FACS (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, COL George Peoples, MD, FACS, Chief, Surgical Oncology, Brooke Army Medical Center; Director and Principal Investigator, Cancer Vaccine Development Program, Walter Reed Army Medical Center
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-20012
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine (Experimental): HLA-A2+ and HLA-A3+ patients are administered the E75+GM-CSF vaccine.
  Interventions: Biological: E75 + GM-CSF vaccine
- Control/observation (No Intervention): HLA-A2- and HLA-A3- patients are prospectively followed for disease recurrence. Control patients are not vaccinated.

INTERVENTIONS:
Biological: E75 + GM-CSF vaccine — The 1 ml by volume vaccine is administered intradermally in 0.5 ml inoculums at two different sites within 5 cm of each other on an extremity. Vaccinations will be given according to the schedule the patient has been assigned and will be administered in the same lymph node draining area (same arm or thigh). In addition, an optional booster inoculation as requested by previously vaccinated patients will be offered every 6 months for the duration of the protocol. The dose will be determined by the PI based on the patient's response to the initial vaccination series.
  Arms: Vaccine

SUMMARY:
The objectives of this study are the following:

1. To assess safety and document local and systemic toxicity to the peptide vaccine (E75) in node-negative breast cancer patients.
2. To determine the optimal dose of the immunoadjuvant, GM-CSF, necessary to elicit an in vivo cellular immune response to the peptide vaccine yet limit toxicity.
3. To determine the optimal inoculation schedule to elicit an in vivo cellular immune response to the peptide vaccine.
4. To correlate the efficiency of eliciting an in vivo cellular immune response to the peptide vaccine with the degree of HER2/neu expression in the patient's tumor.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy and second most common cause of cancer-specific death among women in the United States. Despite advances in the diagnosis and treatment of breast cancer, one third of the women who develop the disease will die of the disease, accounting for approximately 46,300 deaths/year. While good primary therapies are available to treat early stage breast cancer, there is a substantial failure rate to these therapies in more advanced disease.

Advances in the understanding of the immune response to cancer have led to the genesis of immunotherapeutic approaches. Specifically, the development of anti-cancer vaccines holds promise as an adjuvant and preventive therapy for patients after primary surgical and medical treatment for breast cancer, but who are at a high risk for recurrence. While patients with hormone receptor positive tumors have the option to undergo hormonal therapy, recurrence is especially high among estrogen receptor/progesterone receptor (ER/PR) negative patients. For these patients, currently there is no good treatment option after completion of primary therapy; close surveillance and watchful waiting is the standard. It is this population of patients that we have targeted with a vaccine strategy to induce cellular immunity.

In our first vaccine study, (WU # 00-2005: Phase Ib Trial of HER2/neu Peptide (E75) Vaccine in Breast Cancer Patients at High Risk for Recurrence after Surgical and Medical Therapies) we have vaccinated node-positive, HER2/neu-positive breast cancer patients with an immunogenic peptide from the HER2/neu protein mixed with a FDA-approved immunoadjuvant, GM-CSF. The study is still enrolling patients, but to date the vaccine has been safe with very limited toxicity and has been very effective at inducing an immune response to the vaccinated peptide. However, it is too early to determine if this immunity will be protective against disease recurrence.

However, with the early immunologic success of the trial, we now intend to more thoroughly study the optimal dose and schedule of vaccinations necessary to efficiently raise immunity against the peptide. In order to study these permeations, we will need to vaccinate significantly more patients; therefore, we propose to vaccinate node-negative breast patients since 75-80% of patients present with early stage breast cancer. Furthermore, we intend to vaccinate patients regardless of their HER2/neu status in order to determine the impact of prior exposure to this antigen on our ability to raise immunity against HER2/neu. Are patients with prior exposure to HER2/neu sensitized or tolerized to this antigen? This question must be answered in order to determine the usefulness of this vaccine as truly preventive in a cancer-naïve population.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer and negative lymph nodes
2. HLA-A2+ and/or HLA-A3+ to receive the vaccine. HLA-A2-, HLA-A3- patients will be eligible to be included in the control group.
3. Immunologically intact with a good performance status (defined below).
4. Without evidence of disease.
5. Patients may enroll while receiving appropriate hormonal therapy for their disease.
6. Completion of all standard first-line therapies (but may still be on hormonal therapy)

Exclusion Criteria:

1. HLA-A2- and/or HLA-A3- patients will not be vaccinated
2. Anergic by the Mantoux panel of recall antigens
3. Receiving immunosuppressive therapy
4. In poor health (Karnofsky <60%, ECOG >2)
5. Tbili >1.5 mg/dL and creatinine>2 mg/dL
6. Pregnancy (urine HCG)
7. Active metastatic disease
8. Involved in other experimental protocols (unless approval is first obtained by the other study PI)
9. Refusal of standard therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2002-12; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are the safety and optimal dosing of the vaccine to induce an in vivo peptide-specific immune response. | Time period needed to determine the maximum tolerated and optimal biologic doses (30 days after each monthly dose)

SECONDARY OUTCOMES:
Time to recurrence is measured as a secondary outcome measure. | 30 days after each monthly vaccine, then per standard of care for breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, Principal Investigator — Cancer Vaccine Development Program
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Windber Medical Center, Windber, Pennsylvania

REFERENCES:
- [Background] Mittendorf EA, Storrer CE, Shriver CD, Ponniah S, Peoples GE. Investigating the combination of trastuzumab and HER2/neu peptide vaccines for the treatment of breast cancer. Ann Surg Oncol. 2006 Aug;13(8):1085-98. doi: 10.1245/ASO.2006.03.069. Epub 2006 Jul 24. PMID 16865596
- [Background] Dehqanzada ZA, Storrer CE, Hueman MT, Foley RJ, Harris KA, Jama YH, Kao TC, Shriver CD, Ponniah S, Peoples GE. Correlations between serum monocyte chemotactic protein-1 levels, clinical prognostic factors, and HER-2/neu vaccine-related immunity in breast cancer patients. Clin Cancer Res. 2006 Jan 15;12(2):478-86. doi: 10.1158/1078-0432.CCR-05-1425. PMID 16428490
- [Background] Woll MM, Fisher CM, Ryan GB, Gurney JM, Storrer CE, Ioannides CG, Shriver CD, Moul JW, McLeod DG, Ponniah S, Peoples GE. Direct measurement of peptide-specific CD8+ T cells using HLA-A2:Ig dimer for monitoring the in vivo immune response to a HER2/neu vaccine in breast and prostate cancer patients. J Clin Immunol. 2004 Jul;24(4):449-61. doi: 10.1023/B:JOCI.0000029117.10791.98. PMID 15163902
- [Result] Peoples GE, Gurney JM, Hueman MT, Woll MM, Ryan GB, Storrer CE, Fisher C, Shriver CD, Ioannides CG, Ponniah S. Clinical trial results of a HER2/neu (E75) vaccine to prevent recurrence in high-risk breast cancer patients. J Clin Oncol. 2005 Oct 20;23(30):7536-45. doi: 10.1200/JCO.2005.03.047. Epub 2005 Sep 12. PMID 16157940
- [Result] Mittendorf EA, Gurney JM, Storrer CE, Shriver CD, Ponniah S, Peoples GE. Vaccination with a HER2/neu peptide induces intra- and inter-antigenic epitope spreading in patients with early stage breast cancer. Surgery. 2006 Mar;139(3):407-18. doi: 10.1016/j.surg.2005.06.059. PMID 16546506
- [Result] Hueman MT, Stojadinovic A, Storrer CE, Dehqanzada ZA, Gurney JM, Shriver CD, Ponniah S, Peoples GE. Analysis of naive and memory CD4 and CD8 T cell populations in breast cancer patients receiving a HER2/neu peptide (E75) and GM-CSF vaccine. Cancer Immunol Immunother. 2007 Feb;56(2):135-46. doi: 10.1007/s00262-006-0188-9. Epub 2006 Jun 17. PMID 16783576
- [Result] Dehqanzada ZA, Storrer CE, Hueman MT, Foley RJ, Harris KA, Jama YH, Shriver CD, Ponniah S, Peoples GE. Assessing serum cytokine profiles in breast cancer patients receiving a HER2/neu vaccine using Luminex technology. Oncol Rep. 2007 Mar;17(3):687-94. PMID 17273752
- [Result] Stojadinovic A, Mittendorf EA, Holmes JP, Amin A, Hueman MT, Ponniah S, Peoples GE. Quantification and phenotypic characterization of circulating tumor cells for monitoring response to a preventive HER2/neu vaccine-based immunotherapy for breast cancer: a pilot study. Ann Surg Oncol. 2007 Dec;14(12):3359-68. doi: 10.1245/s10434-007-9538-x. Epub 2007 Sep 29. PMID 17906897
- [Result] Peoples GE, Holmes JP, Hueman MT, Mittendorf EA, Amin A, Khoo S, Dehqanzada ZA, Gurney JM, Woll MM, Ryan GB, Storrer CE, Craig D, Ioannides CG, Ponniah S. Combined clinical trial results of a HER2/neu (E75) vaccine for the prevention of recurrence in high-risk breast cancer patients: U.S. Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Clin Cancer Res. 2008 Feb 1;14(3):797-803. doi: 10.1158/1078-0432.CCR-07-1448. PMID 18245541
- [Result] Amin A, Benavides LC, Holmes JP, Gates JD, Carmichael MG, Hueman MT, Mittendorf EA, Storrer CE, Jama YH, Craig D, Stojadinovic A, Ponniah S, Peoples GE. Assessment of immunologic response and recurrence patterns among patients with clinical recurrence after vaccination with a preventive HER2/neu peptide vaccine: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer Immunol Immunother. 2008 Dec;57(12):1817-25. doi: 10.1007/s00262-008-0509-2. Epub 2008 Apr 8. PMID 18392824
- [Result] Mittendorf EA, Holmes JP, Ponniah S, Peoples GE. The E75 HER2/neu peptide vaccine. Cancer Immunol Immunother. 2008 Oct;57(10):1511-21. doi: 10.1007/s00262-008-0540-3. Epub 2008 Jun 7. PMID 18536917
- [Result] Holmes JP, Gates JD, Benavides LC, Hueman MT, Carmichael MG, Patil R, Craig D, Mittendorf EA, Stojadinovic A, Ponniah S, Peoples GE. Optimal dose and schedule of an HER-2/neu (E75) peptide vaccine to prevent breast cancer recurrence: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2008 Oct 1;113(7):1666-75. doi: 10.1002/cncr.23772. PMID 18726994
- [Result] Holmes JP, Clifton GT, Patil R, Benavides LC, Gates JD, Stojadinovic A, Mittendorf EA, Ponniah S, Peoples GE. Use of booster inoculations to sustain the clinical effect of an adjuvant breast cancer vaccine: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2011 Feb 1;117(3):463-71. doi: 10.1002/cncr.25586. Epub 2010 Sep 15. PMID 20845479
- [Result] Patil R, Clifton GT, Holmes JP, Amin A, Carmichael MG, Gates JD, Benavides LH, Hueman MT, Ponniah S, Peoples GE. Clinical and immunologic responses of HLA-A3+ breast cancer patients vaccinated with the HER2/neu-derived peptide vaccine, E75, in a phase I/II clinical trial. J Am Coll Surg. 2010 Feb;210(2):140-7. doi: 10.1016/j.jamcollsurg.2009.10.022. Epub 2009 Dec 22. PMID 20113933
- [Result] Mittendorf EA, Clifton GT, Holmes JP, Clive KS, Patil R, Benavides LC, Gates JD, Sears AK, Stojadinovic A, Ponniah S, Peoples GE. Clinical trial results of the HER-2/neu (E75) vaccine to prevent breast cancer recurrence in high-risk patients: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2012 May 15;118(10):2594-602. doi: 10.1002/cncr.26574. Epub 2011 Oct 11. PMID 21989902
- [Result] Benavides LC, Sears AK, Gates JD, Clifton GT, Clive KS, Carmichael MG, Holmes JP, Mittendorf EA, Ponniah S, Peoples GE. Comparison of different HER2/neu vaccines in adjuvant breast cancer trials: implications for dosing of peptide vaccines. Expert Rev Vaccines. 2011 Feb;10(2):201-10. doi: 10.1586/erv.10.167. PMID 21332269
- [Result] Benavides LC, Gates JD, Carmichael MG, Patil R, Holmes JP, Hueman MT, Mittendorf EA, Craig D, Stojadinovic A, Ponniah S, Peoples GE. The impact of HER2/neu expression level on response to the E75 vaccine: from U.S. Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Clin Cancer Res. 2009 Apr 15;15(8):2895-904. doi: 10.1158/1078-0432.CCR-08-1126. Epub 2009 Apr 7. PMID 19351776
- [Result] Hueman MT, Stojadinovic A, Storrer CE, Foley RJ, Gurney JM, Shriver CD, Ponniah S, Peoples GE. Levels of circulating regulatory CD4+CD25+ T cells are decreased in breast cancer patients after vaccination with a HER2/neu peptide (E75) and GM-CSF vaccine. Breast Cancer Res Treat. 2006 Jul;98(1):17-29. doi: 10.1007/s10549-005-9108-5. Epub 2006 Jun 7. PMID 16758122